CLINICAL TRIAL: NCT01253915
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of Nasal Carbon Dioxide in the Treatment of Moderate to Severe Migraine
Brief Title: The Effect of Nasal Carbon Dioxide in the Treatment of Moderate to Severe Migraine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment and lack of funding for study
Sponsor: Capnia, Inc. (Industry)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency); United States Naval Medical Center, Portsmouth (U.S. Federal Agency); Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C113
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbon Dioxide (Experimental)
  Interventions: Drug: Nasal Carbon Dioxide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nasal Carbon Dioxide — 10 sec/nostril up to 4 times to treat one migraine
  Arms: Carbon Dioxide
Drug: Placebo — 10 sec/nostril up to 4 times to treat a migraine
  Arms: Placebo

SUMMARY:
This multi-center, double-blind, placebo-controlled, parallel group trial carbon dioxide in the treatment of moderate to severe migraine. At approximately 8 US sites, approximately 450 patients who meet the eligibility criteria will be randomized to active or placebo in a 1:1 ratio to ensure that 400 patients will treat at least one moderate to severe migraine with the study drug.

Patients will be randomized to one of two treatment groups and be provided with either an active or placebo dispenser.

All patients will administer study drug for 10 seconds to each nostril when experiencing a qualifying headache. Patients will assess their pain and other migraine-related symptoms in a patient diary. If a patient still has pain and/or any other symptoms after the initial dose then the patient may opt to take 3 more doses to treat the headache.

Each patient's participation in the study may last up to 56 days or once the patient treats 4 headaches with the study drug, whichever occurs first.

There will be a total of 2 scheduled clinic visits:

* Visit 1 Screening/Randomization
* Visit 2 End of Study (within 7 days after the patients treats his/her fourth headache or after the end of the 56-day treatment period, whichever occurs first)

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand informed consent form and voluntarily consent to participate in this study by signing the IRB-approved informed consent form
* Males and females ages 18 - 65 years
* Established diagnosis of migraine with or without aura per ICHD-II (patients with a diagnosis of only menstrual migraine are not eligible)
* At least a one-year history of migraine symptoms with or without aura
* Age at migraine onset less than 50 years
* History of 2-8 migraine attacks per month during the 3 months prior to randomization
* Females of childbearing potential must commit to using an acceptable method of birth control (e.g., oral birth control pills, intrauterine device (IUD), or a double-barrier method of contraception) through 7 days after last study drug administration. To be considered not of childbearing potential, females must be post-menopausal for at least 2 years or be surgically sterile

Exclusion Criteria:

* Have less than 48 hours of freedom from headache between attacks of migraine
* Have 15 or more headache days per month
* Have migraine secondary to traumatic brain injury (TBI)
* Are unable to comply with protocol requirements
* Females who are pregnant or breast-feeding and/or plan to become pregnant or to breast-feed during study participation or within 7 days after last study drug administration
* Have changed their usage of prescription migraine prophylaxis medications within 12 weeks prior to randomization
* Use antipsychotic or antidepressant medications (unless only for migraine prophylaxis) within 12 weeks prior to randomization and for the duration of the study
* Have a history of alcohol or drug abuse within 2 years prior to randomization
* Have a psychiatric disease which may prevent patient compliance or otherwise interfere with the ability of the patient to participate in the study
* Have a medical condition that makes study participation unwise in the opinion of the Investigator (e.g., significant COPD, heart disease, etc.)
* Have a concurrent diagnosis of temporomandibular disorders (TMD) or trigeminal neuralgia requiring treatment
* Clinically significant deviated septum, nasal polyps or other nasal condition that prevents unrestricted breathing through each nostril
* Are going to travel extensively by airplane during the 56-day treatment period (e.g., anticipated travel by airplane more than 25% of the 56-day treatment period, 14 days)
* Have a member of the same household also participating in this study
* Use of any investigational or experimental therapy within 30 days of randomization
* Have participated in another study with nasal CO2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who are pain-free | at 2 hours after study drug administration

SECONDARY OUTCOMES:
The proportion of patients who are nausea/vomiting free | at 2 hours after study drug administration
The proportion of patients who are phonophobia free | at 2 hours after study drug administration
The proportion of patients who are photophobia free | at 2 hours after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Bertrand, DDS, Study Chair — National Naval Medical Center, Bethesda
Locations (3):
- United States (3):
  - Naval Medical Center San Diego - Dept of Neurology, San Diego, California
  - Walter Reed National Military Medical Center - Dept of Neurology, Bethesda, Maryland
  - Naval Medical Center Portsmouth - Dept of Neurology, Portsmouth, Virginia